CLINICAL TRIAL: NCT00077090
Title: Randomized Phase II Trial Of Hyperbaric Oxygen Therapy In Patients With Chronic Arm Lymphoedema After Radiotherapy For Cancer
Brief Title: Hyperbaric Oxygen Therapy Compared With Standard Therapy in Treating Chronic Arm Lymphedema in Patients Who Have Undergone Radiation Therapy for Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000349496; RMNHS-HOT; EU-20337
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer; Lymphedema; Perioperative/Postoperative Complications; Radiation Fibrosis
Keywords: lymphedema; radiation fibrosis; perioperative/postoperative complications; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Postoperative Complications; Radiation Fibrosis Syndrome | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Drug: hyperbaric oxygen

SUMMARY:
RATIONALE: Hyperbaric oxygen therapy may be effective in repairing damaged tissue and reducing lymphedema caused by radiation therapy for cancer.

PURPOSE: This randomized phase II trial is studying hyperbaric oxygen to see how well it works compared to standard therapy in treating chronic arm lymphedema in patients who have undergone radiation therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of hyperbaric oxygen (HBO) therapy vs standard management, in terms of reduction of lymphedema, in patients with chronic arm lymphedema after radiotherapy for cancer.

Secondary

* Determine the mechanisms of tissue reperfusion and healing in patients treated with HBO therapy.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo hyperbaric oxygen therapy over 90 minutes 5 days a week for 6 weeks.
* Arm II: Patients receive standard management. Patients are followed at 3, 6, 9, 12, and 15 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 63 patients (42 for arm I and 21 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of early breast cancer (T1-3, N0-1, M0)
* Prior breast surgery with or without axillary dissection
* Prior breast/chest wall radiotherapy with or without radiotherapy to the supraclavicular fossa and/or axilla, completed at least 2 years ago
* Arm lymphedema

  * At least 15% increase in arm volume
* No evidence of cancer recurrence
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Female or male

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No chronic obstructive airway disease
* No bullous lung disease
* No acute or chronic pulmonary infection
* No uncontrolled asthma
* No untreated pneumothorax

Other

* Physically and psychologically fit for HBO therapy
* No claustrophobia
* No epilepsy
* No eustachian tube dysfunction
* No recurrent attacks of vertigo
* No contraindication to MRI (e.g., intracranial ferrous material)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* No prior ear operations

Other

* No prior hyperbaric oxygen (HBO) therapy, except as treatment for decompression illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
Volume of the affected limb, expressed as a percentage of the contralateral limb Volume on the day of measurement, as measured by perometer 12 months after baseline assessment

SECONDARY OUTCOMES:
Patient self-assessments, using specific quality of life scale in upper limb lymphoedema and the UK SF-36 Health Survey Questionnaire, at 3, 6, 9 and 12 months after baseline assessment
99Tc-nanocolloid clearance rate as measured by quantitative lymphoscintigraphy 12 months after baseline assessment
Extracellular water content as measured by EdemaMeter (bioimpedance measurements) 12 months after baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Royal Hospital Haslar, Gosport, England
  - Hull Royal Infirmary, Hull, England
  - London Hyperbaric Medicine Limited at Whipps Cross Hospital, London, England
  - Diving Diseases Research Centre, Plymouth, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England